CLINICAL TRIAL: NCT05711186
Title: Structured Shared Decision Making for Patients Undergoing Elective Surgical or Transcatheter Aortic Valve Replacement (TOGETHER): A Randomized-controlled Trial
Brief Title: Structured Shared Decision Making for Patients Undergoing SAVR or TAVR
Acronym: TOGETHER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TOGETHER (2022-01691)
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Aortic Valve Stenosis; Symptomatic Aortic Stenosis
Keywords: Symptomatic Aortic Stenosis; Aortic Valve Stenosis; SAVR (Surgical Aortic Valve Replacement); Shared Decision-Making; TAVR (Transcatheter Aortic Valve Replacement); TAVI (Transcatheter Aortic Valve Implantation); Decision Support Techniques
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured SDM (Other): Structured shared decision making for the choice between SAVR and TAVR
  Interventions: Other: Structured SDM
- Usual Care (Other): Usual care for the choice between SAVR and TAVR
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Structured SDM — The conversation between the heart team member and the patient will be structured according the adapted three-talk model for patients with symptomatic aortic stenosis and using the American College of Cardiology's decision aid for patients deciding between TAVR and SAVR
  Arms: Structured SDM
Other: Usual Care — Usual care will include baseline visits without a structured SDM approach. Usual care includes at least one decision making talk with a heart team member discussing information about the disease, treatment options as well as benefits and risks of each procedure.
  Arms: Usual Care

SUMMARY:
Transcatheter aortic valve replacement (TAVR) is a well-established alternative to surgical aortic valve replacement (SAVR) for the treatment of patients with severe aortic stenosis regardless of surgical risk. While TAVR and SAVR share some of the benefits and risks, they importantly differ with regards to invasiveness, time to recovery, hemodynamics, as well as options for re-intervention and possibly valve durability. An early benefit of TAVR may be offset by late risks. Therefore, current guidelines of the European Society of Cardiology recommend an integration of patient values and preferences for the selection of the treatment modality.

The objective of the TOGETHER trial is to investigate the efficacy of a structured shared decision making approach (SDM) to improve patient-centered outcomes for the choice between SAVR and TAVR.

TOGETHER is an investigator-initiated, randomized, open-label, single-center clinical trial. A total of 140 patients referred for treatment of symptomatic severe aortic stenosis and deemed to undergo TAVR or SAVR according to heart team decision will be randomized in a 1:1 ratio to structured SDM or usual care.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years
2. Symptomatic severe aortic stenosis defined by an aortic valve area ≤1.0 cm2 or an aortic valve area indexed to body surface area <0.6cm2/m2
3. Both SAVR and transfemoral TAVR as reasonable treatment options based on heart team decision

Exclusion Criteria:

1. Life expectancy <1 year irrespective of valvular heart disease
2. Inability to provide informed consent
3. Participation in another clinical trial with an active intervention

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Patient decisional conflict | 3 days post baseline visit
  Assessed by decisional conflict scale (ranges from 0 to 100, with higher scores indicating a worse outcome)
Patient decisional regret | 30 days post TAVR/SAVR
  Assessed by the decision regret scale (ranges from 0 to 100, with higher scores indicating a worse outcome)

SECONDARY OUTCOMES:
Patient-centered communication | 3 days post baseline visit
  Assessed by CollaboRATE scale (ranges from 0 to 100, with higher scores indicating a better outcome)
Patient knowledge about the treatment options and outcomes | 3 days post baseline visit
  Assessed by 6 multiple-choice items (ranges from 0 to 6, with higher scores indicating a better outcome)
Patient procedural satisfaction | 3 days post baseline visit
  Assessed by Likert Scale (ranges from 1 to 5, with higher scores indicating a better outcome)
Patient decisional satisfaction | 3 days post baseline visit; 30 days and 1 year post TAVR/SAVR
  Assessed by Likert Scale (ranges from 1 to 5, with higher scores indicating a better outcome)
Incorporation of patient values | 3 days post baseline visit
  Assessed by values clarity subscore of the decisional conflict scale (ranges from 0 to 100, with higher scores indicating a worse outcome)
Patient feeling of not being informed | 3 days post baseline visit
  Assessed by informed subscore of the decisional conflict scale (ranges from 0 to 100, with higher scores indicating a worse outcome)
Quality of choice | 3 days post baseline visit
  Assessed by effective decision subscore of the decisional conflict scale (ranges from 0 to 100, with higher scores indicating a worse outcome)
Patient decisional regret | 1 year post TAVR/SAVR
  Assessed by the decision regret scale (ranges from 0 to 100, with higher scores indicating a worse outcome)
Patient health-related quality of life | 30 days post TAVR/SAVR
  Assessed by KCCQ 12 (Kansas City Cardiomyopathy Questionnaire) (ranges from 0 to 100, with higher scores indicating a better outcome)
The proportion of patients choosing TAVR/SAVR | Baseline
  Number of participants choosing valve replacement by TAVR or SAVR
The incidences of major clinical adverse events | 30 days and 1 year post TAVR/SAVR
  All-cause mortality, stroke, transient ischemic attack, bleeding event, kidney injury, systemic embolism, myocardial infarction, new onset atrial fibrillation, permanent pacemaker implantation and intervention related to the device

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Pilgrim, Prof., Principal Investigator — Department of Cardiology, University Hospital Bern, Inselspital, Bern; Christoph Ryffel, Dr. med., Principal Investigator — Department of Cardiology, University Hospital Bern, Inselspital, Bern
Locations (1):
- Bern University Hospital, Dep. of Cardiology, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No